CLINICAL TRIAL: NCT06182215
Title: Postoperative Neurocognitive Dysfunction After Major Abdominal Surgery: A Prospective Observational Cohort Study
Brief Title: PostoperAtive Neurocognitive Dysfunction After Major AbdomiNal Surgery (PANDAMAN)
Acronym: PANDAMAN
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2023-143-v2
Record Dates: First submitted 2023-12-02; First posted 2023-12-26 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Elective Major Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective observational cohorts: patients undergoing elective major abdominal surgery (estimated operation time over 2 hours)

SUMMARY:
Predisposing and precipitating factors for perioperative delirium for the elderly remain elusive. This research will be conducted to determine risk factors of postoperative delirium.

DETAILED DESCRIPTION:
This study intends to include 500 participants over 65 years old undergoing elective abdominal major surgery. The primary outcome is incidence of delirium at 7 days postoperatively, and the secondary outcomes include preoperative sleep disorders(Athens In-somnia Scale, AIS), postoperative cognitive impairment (Abbreviated Mental Test Score, AMTS), postoperative pain (NRS pain score), incidence of significant postoperative complications, length of hospital stay, and serum biomarkers levels.

ELIGIBILITY:
Inclusion Criteria:

1. 65 to 90 years old to receive elective major abdominal surgery (expected operation time over 2 hours); ,
2. American society of Aneshesiologists（ASA）physical status I-III;

Exclusion Criteria:

1. Mini-Mental State Examination (MMES) score < 15;
2. Renal failure (requiring dialysis) or liver failure (Child-Pugh score > 5);
3. Severe impairment due to structural or hypoxic brain injury, more than 2 days in ICU one month before surgery;
4. Underwent major heart, lung or abdominal surgery within 1 year;
5. Positive for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) or symptomatic (e.g. fever, cough, loss of taste/smell);
6. The cognitive assessment cannot be completed because the subject is blind, deaf, or unable to communicate in the local language;
7. Long-term follow-up unavailable (homelessness, active psychosis or substance abuse).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 to 90 years who received elective major abdominal surgery (estimated operation time over 2 hours)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium during first 7 days after surgery | Consecutive 7 days after the surgery or hospital discharge, whichever comes first.
  The result of 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) is positive.

SECONDARY OUTCOMES:
Preoperative cognitive function | Day 1 before surgery
  The Mini-Mental State Examination scale will be used to assist in evaluating preoperative cognitive function in patients. The scale's testing items include orientation, memory, calculation, language, visual space, use, and attention, with a total score of 30. The higher the score, the better the cognitive function, and the score below 27 indicates possible cognitive impairment.
Age-adjusted Charlson Comorbidity Index | Day 1 before surgery
  Age-adjusted Charlson Comorbidity Index is a method used to evaluate the impact of multiple diseases on a patient's health status. The scale includes a total of 16 common co-morbidity diseases, which is divided into 4 categories according to different disease severity, with scores of 1,2,3 or 6. The higher the score, the more kinds of diseases the patient suffers at the same time, and their health status may be more complex and fragile.
Preoperative anxiety | Day 1 before surgery, day 3 after surgery
  Hamilton Anxiety Scale will be used to evaluate the patient's anxiety status, which consist of 14 items. All items are scored on a 5-level scale of 0-4, with criteria for each level being none, mild, moderate, severe, and extremely severe. The higher the score, the more severe the anxiety symptoms.
Serum biomakers levels | Within 15 minutes after induction of anesthesia, day 3 after surgery
  Extract venous blood samples from the target patient, store and centrifuge the Samples appropriately. Quantitatively detect the serum biomakers levels, such as NFL, using enzyme-linked immunosorbent assay, and retest the concentration changes of these biomarkers 3 days after surgery.
Preoperative Sleep quality | Day 1 before surgery, Day 3 after surgery
  Athens Insomnia Scale will be used to assess the patient's preoperative sleep quality. A maximum total score of 24 indicates the most severe symptoms of insomnia, while a cut-off point of ≥6 represents a minimum criterion for the confirmation of insomnia symptoms.
Postoperative pain | Consecutive 7 days after the surgery or hospital discharge, whichever comes first.
  Postoperative pain will be evaluated by Number Rating Scale, which is composed of 11 numbers from 0 to 10, where 0 is no pain or hurt and 10 is the most or worst pain. The higher the number, the more severe the pain.
Length of hospital stay | Up to 24 weeks after surgery
  The length of patient hospital stay will be supplemented through Hospital Information System after surgery.
Health status and quality of life | Day 1 before surgery, day 30 after surgery
  Short Form 36 Health Survey will be used to estimate the health status and quality of life of patients. This scale includes 8 dimensions and a total of 36 questions, convert the scores of each section into a range of 0 to 100, where 100 represents the "best health state", and the lower the score, the worse the health condition.
Postoperative adverse complications | Up to day 30 after surgery
  Include but limited to hospital readmissions 30 days after surgery, unplaned reoperations, stroke, kidney failure, and wound infections.
All-cause mortality at 30 days after surgery | Up to day 30 after surgery
  The ratio of total deaths from all causes to the population.
Postoperative cognitive dysfunction | Day 1 before surgery, day 30 after surgery, day 90 after surgery
  The Abbreviated Mental Test Score will be administered by telephone respectively 1 month and 3 months after surgery to identify long-term cognitive consequences of anaesthesia and postoperative delirium. The scale consists of 10 questions with a total of 10 points, the higher the score, the better the cognitive function, and those with score < 8 will be identified as possible neurocognitive dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PhD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yet-set University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen H, Ding M, Ma X, Deng W, Liang B, Ruan X, Zhang X. The multidimensional physiological, psychological, and social influencing factors of perioperative neurocognitive disorders in elderly Chinese patients undergoing major abdominal surgery: study protocol of a prospective cohort study. BMC Geriatr. 2026 Feb 2. doi: 10.1186/s12877-026-07052-2. Online ahead of print. PMID 41629790